CLINICAL TRIAL: NCT05548218
Title: Care Companion: A Pragmatic Trial Conducting Automated Health Educations Among Patient With Type-2 Diabetes Utilizing a Digital Health Pathway
Brief Title: Care Companion Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Nirav Shah, Medical Director of Quality Innovation and Clinical Practice Analytics, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EH22-331
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- New diagnosis of diabetes control group (No Intervention)
- New diagnosis of diabetes intervention group (Experimental)
  Interventions: Other: Automated health education using a digital health pathway
- Uncontrolled diabetes control group (No Intervention)
- Uncontrolled diabetes intervention group (Experimental)
  Interventions: Other: Automated health education using a digital health pathway

INTERVENTIONS:
Other: Automated health education using a digital health pathway — MyChart Care Companion is an interactive, individualized plan of care delivered to at-risk patients through user-friendly, accessible technology. Care Companion is a digital health pathway housed within EPIC. Care Companion features are integrated into the existing MyChart mobile app, which is part of Epic, and is available for iOS and Android devices. The interactive plan of care delivers notifications to patients' phones, prompts patients to complete educational session in the mobile app, analyzes questionnaire responses and patient-reported data, and orchestrates changes to the plan and escalations as needed to help patients, their caregivers, and care managers stay on top of the patient care. In addition to mobile phone, patients can also now access MyChart Care Companion on webpages via computers. The automated pathway assigns patient interactive health education materials during the study.
  Arms: New diagnosis of diabetes intervention group; Uncontrolled diabetes intervention group

SUMMARY:
Digital health interventions have the potential to help patients with diabetes effectively manage their disease at home. Many digital health studies provide patients with educational materials and self-care recommendations. The digital health interventions allow patients to conveniently access these materials on their phones or computers, and enable care teams to provide essential knowledge for diabetes management. Digital health based education intervention is a reasonably inexpensive method that offers high coverage and motivational encouragement to help patients improve their health at home.This study aims to provide patients with timely education for diabetes management and has the potential to improve clinical outcomes for patients with diabetes.

DETAILED DESCRIPTION:
This study is a prospective, randomized control, pragmatic trial of patients with diabetes, including patients newly diagnosed with diabetes and patients with uncontrolled diabetes. This study focuses on delivering educational materials through the MyChart Care Companion pathway to conduct timely educations and assess patient medication adherence level and activity level. This is a minimal risk study without intervention procedures.

There are two Type 2 Diabetes subjects groups uncontrolled diabetes and new diabetics. Each group will be randomized 1 to 1 to either the Care Companion program or control group which receives a one-page document on diabetic care. The Care Companion program is a digital interactive weekly program that includes modules on health and nutrition education and weekly activity and medication adherence check-ins. There are weekly modules that are completed over 16 weeks.

The objective is to provide timely education to patients with type 2 diabetes through MyChart Care Companion pathway, with the aim of improving patient's self management knowledge. We will also evaluate patient experience and acceptance of the MyChart Care Companion features.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new type 2 diabetes diagnosis within 1 year at time of enrollment and has an A1c level over 6.5%, or patients with a type 2 diabetes diagnosis over an year and has an A1c level over 8% at time of enrollment
* Patient able to speak and understand English
* Patient is at least 18 years of age

Exclusion Criteria:

* Patient has cognitive limitations that, in the opinion of their provider, limit the patient's ability to understand study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in A1C level | 16 weeks
  Our primary clinical outcome of interest would be the change in A1c levels measured at baseline during enrollment and at the 12-16 week mark of the study.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Swedish Covenant Hospital, Chicago, Illinois
  - NorthShore University HealthSystem Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem HighlandPark Hospital, Highland Park, Illinois

IPD SHARING:
Plan to Share IPD: No